CLINICAL TRIAL: NCT02704624
Title: The Impact of Serum Vitamin D and Calcium Levels on the Body Composition, Bone Mineral Density, Muscle Strength, Exercise Tolerance, Fatigue and Inflammatory Activity in Patients With Crohn's Disease: a Randomized Controlled Trial
Brief Title: Effects of Supplementation of Vitamin D in Patients With Crohn's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of Juiz de Fora (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Lorena Nagme de Oliveira Pinto, lecturer, Federal University of Juiz de Fora
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE41674814500005147
Record Dates: First submitted 2016-02-24; First posted 2016-03-10 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-04

CONDITIONS: Crohn Disease; Vitamin D Deficiency; Fatigue; Sarcopenia; Muscle Weakness; Disorder of Bone Density and Structure, Unspecified
Keywords: Crohn Disease; Fatigue; Osteopenia; Exercise Tolerance; Vitamin d
MeSH Terms: conditions — Crohn Disease; Vitamin D Deficiency; Fatigue; Sarcopenia; Muscle Weakness; Bone Diseases, Metabolic | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, placebo-controlled study will be performed. After the evaluation of serum vitamin D levels, patients with vitamin D below 30ng/mL will be randomized into two groups. One group will receive supplementation with cholecalciferol (vitamin D3) tablets and the other group will receive placebo. Those will be provided at no cost to the patients. The dosage of 1.500-2.000 IU (International Units) vitamin D/day is recommended in order to meet the need of vitamin D above 30ng/mL in adults. However, a dose at least 2 to 3 times higher is recommended for CD patients due to malabsorption, significant loss of adipose tissue and use of glucocorticoids. Thus, the dose of 50,000IU/week will be administered in a single dose. The patients drawn to the placebo group will receive inert content tablets without therapeutic effect. After the study completion, these control patients will receive complete treatment for hypovitaminosis D.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the pharmacist responsible for confection of the tablets will know who will receive vitamin d or placebo, according to a list of randimization generated in the computer by the statistician. The list will be kept with the pharmacist throughout the intervention.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator): Tablets with 50000UI cholecalciferol (vitamin D3) will be administered, weekly, for six months.
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): The patients selected to the placebo group will receive inert content tablets without therapeutic effect, weekly, for six months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — investigate the relationship between musculoskeletal manifestations, in Crohn population, and the hypovitaminosis D
  Arms: Vitamin D
Other: Placebo — compare the musculoskeletal manifestations of the Placebo group with the group receiving Vitamin D
  Arms: Placebo

SUMMARY:
Thus, the aim of the current study is to assess the influence of vitamin D deficiency and, consequently, of serum calcium deficiency in the body composition, muscular activity, bone mineral density, fatigue, and exercise tolerance of CD patients. Secondly, it also aims to determine the impact of vitamin D supplementation on this population.

DETAILED DESCRIPTION:
This will be a clinical, randomized, controlled, and double-blind trial comprising a consecutive sample of 110 CD patients in remission and low serum vitamin D levels treated by the Gastroenterology team of the Inflammatory Intestinal Disease Clinic at the University Hospital (HU/CAS), Federal University of Juiz de Fora (UFJF). These patients will be divided into two groups with 55 patients each. One group will receive vitamin D supplementation (50.000 UI/week) and the other will receive placebo. Upon the approval by the Ethics Committee of the UFJF, the study aims and procedures will be previously explained to the individuals, who will sign an informed consent form.

The sample size was based on the handgrip strength test, assuming an alpha risk of 5 % and beta risk of 80 %, standard deviation of 2.5, and a difference in magnitude of 30% of response between intervention and placebo group, the sample size needed was 45 patients in each group. Therefore, considering potential losses, 55 patients will be recruited for each group, requiring a total of 110 volunteers.

Study procedure

Phase 1. Assessment All patients in the study will be subjected to the following tests: a. clinical assessment; B. biochemical assessment; c. body composition assessment/anthropometry; d. bone mineral density assessment; e. peripheral muscle strength assessment; f. fatigue assessment; g.Exercise Tolerance Testing

Clinical Assessment of the Disease The following data will be collected in the initial assessment: age, gender, CD duration, data related to the Montreal Classification (age at the time of diagnosis, disease behavior and location), glucocorticoid use and number of exacerbations in the previous year. The inflammatory activity assessment will be held according to the Harvey-Bradshaw Index, When the score is less than 5, the disease is considered to be inactive.

Biochemical Assessment The participants will be instructed to fast 12 hours prior to the blood sampling for analysis. A 5 ml venous blood sample will be collected from the patients in order to determine biochemical parameters. The University Hospital routine laboratory will analyze the venous blood, the levels of C-reactive protein (CRP), calcium, 25-hydroxyvitamin D, parathyroid hormone (PTH) and inflammatory cytokines such as Interleukins (IL) 17, IL 6 and Tumor necrosis factor alfa (TNF-α) . CRP and serum calcium are routinely evaluated in all CD patients under follow-up in the inflammatory bowel disease clinic at HU/CAS.

The following reference values will be taken into consideration regarding 25-hydroxyvitamin D: < 20ng/mL = deficiency, between 21 and 29 ng/mL = insufficiency, and > 30 ng/mL = satisfactory.

Bone Mineral Density Assessment A bone densitometer, Lunar Prodigy Primo (pr + 351035), will be used to measure the patients' bone mineral density (BMD), expressed in g/cm2, by dual-energy x-ray absorptiometry (DXA). The double-energy X-ray densitometry of the skeleton or specific sites such as the spine and the hip is based on the X-rays absorption by the calcium crystals in the bone. The lumbar spine regions between L1 and L4 and those of the total proximal femur will be assessed. The examination will be held under appropriate conditions, according to the technical quality controls. The coefficient of variation for the lumbar spine and total proximal femur will be obtained based on these results. The low BMD will be defined by the reduction greater than -2.0 standard deviations from the reference value mean of healthy individuals, adjusted according to height, age and gender (Z score), in compliance with the official positions of the International Society for Clinical Densitometry (ISCD).

Body Composition Assessment/Anthropometry The assessment will be held through the Quantum BIA (bioelectrical impedance analysis) bioimpedance device. The device is four-pole, has digital display, and provides resistance and reactance values. Total and segmental body composition parameters will be also assessed by DXA expressed in kg.

Muscle Strength Assessment The peripheral muscle strength will be assessed through the maximum voluntary handgrip strength using hand-held dynamometry (HHD), which consists of a simple and objective test that estimates the skeletal muscle function. The Jamar's hydraulic dynamometer will be used, since it is recommended by the American Society of Hand Therapists (ASHT) and is considered the most accurate and precise instrument used to assess HHD .

Fatigue Assessment The questionnaire by Chalder et al. (Annex), which was validated in Brazil will be applied to assess fatigue.

Exercise Tolerance Testing The exercise capacity is assessed by the walking test with progressive loading or Shuttle Walk Test.

Phase 2. Intervention A double-blind, randomized, placebo-controlled study will be performed. After the evaluation of serum vitamin D levels, patients with vitamin D below 30ng/mL will be randomized into two groups. One group will receive supplementation with cholecalciferol (vitamin D3) tablets and the other group will receive placebo. Those will be provided at no cost to the patients. The dosage of 1.500-2.000 IU (International Units) vitamin D/day is recommended in order to meet the need of vitamin D above 30ng/mL in adults. However, a dose at least 2 to 3 times higher is recommended for CD patients due to malabsorption, significant loss of adipose tissue and use of glucocorticoids. Thus, the dose of 50,000IU/week will be administered in a single dose.

The contraindications and precautions on the use of vitamin D will be respected, namely: hypersensitivity to the D-group vitamins, hypercalcemia, hypercalciuria and metastatic calcification; and interactions with digitalis, thiazides, and anticonvulsant and antacid medications.

Despite the possible interference of the skin melanin concentration in vitamin D absorption, no evidence was found to support the differentiated supplementation between Afro descendant and Caucasian individuals.

The patients drawn to the placebo group will receive inert content tablets without therapeutic effect. After the study completion, these control patients will receive complete treatment for hypovitaminosis D.

Throughout the intervention phase, both the treated group and the control group patients will be monitored by phone every 15 days in order to optimize their adhesion.

Phase 3. Reassessment At the end of 6 months of supplementation with cholecalciferol (vitamin D3), this subgroup of patients will be subjected to the same assessments performed in phase 1.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Crohn's Disease (moderate to severe)
* Remission of Crohn's activity
* Reduced blood levels of vitamin D

Exclusion Criteria:

* Presence of other chronic concomitant disease
* Presence of other autoimmune disease
* Presence of sleep disturbance
* Abuse of alcohol and other drugs
* Pregnancy or lactation, climacteric and/or menopausal women
* Adherence to extreme diet (e.g. macrobiotic or vegetarian diet)
* Celiac disease
* Presence of extensive resection of the small intestine (more than 100cm²)
* Patients undergoing vitamin D replacement for the last 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Increase in the grip strength in patients with Crohn under vitamin D supplementation | After 6 months of supplementation with vitamin D
  Grip strength will be expressed in kg

SECONDARY OUTCOMES:
Increase in mineral bone density (MBD) | After 6 months of supplementation with vitamin D
  MBD assessed by DXA, expressed in gr/cm²
Decrease in fecal Calprotectin levels | After 6 months of supplementation with vitamin D
  Levels of calprotectin under 200µg/g
Global reduction in laboratorial inflammatory biomarkers (TNF-α) | After 6 months of supplementation with vitamin D
  TNF-α expressed in pg/ml
Increase in exercise capacity assessed by Shuttle Walk Test (SWT) | After 6 months of supplementation with vitamin D
  Improvement in the distance achieved in the SWT expressed in meters (m)
Increase in lean body mass in patients with Crohn under vitamin D supplementation | After 6 months of supplementation with vitamin D
  Body mass will be assessed by DXA and will be expressed in kg
Reduction in fatigue perception in patients with Crohn under vitamin D supplementation | After 6 months of supplementation with vitamin D
  Fatigue will be measured by the Chalder Fatigue Questionnaire (CFQ). The CFQ is analyzed by 2 domains physical and mental (cutoff: patient's total score higher than 2)
Global reduction in laboratorial inflammatory biomarkers (IL 6) | After 6 months of supplementation with vitamin D
  IL 6 expressed in pg/ml
Global reduction in laboratorial inflammatory biomarkers (IL 17) | After 6 months of supplementation with vitamin D
  IL 17 expressed in pg/ml
Global reduction in laboratorial inflammatory biomarkers (CRP) | After 6 months of supplementation with vitamin D
  CRP expressed in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Júlio MF Chebli, Professor, Principal Investigator — Federal University of Juiz de Fora
Locations (1):
- Universidade Federal de Juiz de Fora, Juiz de Fora, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernstein CN, Seeger LL, Sayre JW, Anton PA, Artinian L, Shanahan F. Decreased bone density in inflammatory bowel disease is related to corticosteroid use and not disease diagnosis. J Bone Miner Res. 1995 Feb;10(2):250-6. doi: 10.1002/jbmr.5650100211. PMID 7754804
- [Background] Beck A, Bager P, Jensen PE, Dahlerup JF. How fatigue is experienced and handled by female outpatients with inflammatory bowel disease. Gastroenterol Res Pract. 2013;2013:153818. doi: 10.1155/2013/153818. Epub 2013 Sep 1. PMID 24072994
- [Background] Cho HJ, Costa E, Menezes PR, Chalder T, Bhugra D, Wessely S. Cross-cultural validation of the Chalder Fatigue Questionnaire in Brazilian primary care. J Psychosom Res. 2007 Mar;62(3):301-4. doi: 10.1016/j.jpsychores.2006.10.018. PMID 17324680
- [Background] Dusso AS, Brown AJ, Slatopolsky E. Vitamin D. Am J Physiol Renal Physiol. 2005 Jul;289(1):F8-28. doi: 10.1152/ajprenal.00336.2004. PMID 15951480
- [Background] Farraye FA, Nimitphong H, Stucchi A, Dendrinos K, Boulanger AB, Vijjeswarapu A, Tanennbaum A, Biancuzzo R, Chen TC, Holick MF. Use of a novel vitamin D bioavailability test demonstrates that vitamin D absorption is decreased in patients with quiescent Crohn's disease. Inflamm Bowel Dis. 2011 Oct;17(10):2116-21. doi: 10.1002/ibd.21595. Epub 2011 Jan 6. PMID 21910173
- [Background] Gaburri PD, Chebli JM, de Castro LE, Ferreira JO, Lopes MH, Ribeiro AM, Alves RA, Froede EC, de Oliveira KS, Gaburri AK, Gaburri D, Meirelles GS, de Souza AF. [Epidemiology, clinical features and clinical course of Crohn's disease: a study of 60 cases]. Arq Gastroenterol. 1998 Oct-Dec;35(4):240-6. Portuguese. PMID 10347705
- [Background] Hwang C, Ross V, Mahadevan U. Micronutrient deficiencies in inflammatory bowel disease: from A to zinc. Inflamm Bowel Dis. 2012 Oct;18(10):1961-81. doi: 10.1002/ibd.22906. Epub 2012 Apr 5. PMID 22488830
- [Background] Iijima H, Shinzaki S, Takehara T. The importance of vitamins D and K for the bone health and immune function in inflammatory bowel disease. Curr Opin Clin Nutr Metab Care. 2012 Nov;15(6):635-40. doi: 10.1097/MCO.0b013e328357f623. PMID 22914505
- [Background] Kim YG, Jang BI. The role of colonoscopy in inflammatory bowel disease. Clin Endosc. 2013 Jul;46(4):317-20. doi: 10.5946/ce.2013.46.4.317. Epub 2013 Jul 31. PMID 23964327
- [Background] van Langenberg DR, Gibson PR. Factors associated with physical and cognitive fatigue in patients with Crohn's disease: a cross-sectional and longitudinal study. Inflamm Bowel Dis. 2014 Jan;20(1):115-25. doi: 10.1097/01.MIB.0000437614.91258.70. PMID 24297056
- [Background] Peyrin-Biroulet L, Fiorino G, Buisson A, Danese S. First-line therapy in adult Crohn's disease: who should receive anti-TNF agents? Nat Rev Gastroenterol Hepatol. 2013 Jun;10(6):345-51. doi: 10.1038/nrgastro.2013.31. Epub 2013 Mar 5. PMID 23458890
- [Background] Pludowski P, Karczmarewicz E, Bayer M, Carter G, Chlebna-Sokol D, Czech-Kowalska J, Debski R, Decsi T, Dobrzanska A, Franek E, Gluszko P, Grant WB, Holick MF, Yankovskaya L, Konstantynowicz J, Ksiazyk JB, Ksiezopolska-Orlowska K, Lewinski A, Litwin M, Lohner S, Lorenc RS, Lukaszkiewicz J, Marcinowska-Suchowierska E, Milewicz A, Misiorowski W, Nowicki M, Povoroznyuk V, Rozentryt P, Rudenka E, Shoenfeld Y, Socha P, Solnica B, Szalecki M, Talalaj M, Varbiro S, Zmijewski MA. Practical guidelines for the supplementation of vitamin D and the treatment of deficits in Central Europe - recommended vitamin D intakes in the general population and groups at risk of vitamin D deficiency. Endokrynol Pol. 2013;64(4):319-27. doi: 10.5603/ep.2013.0012. PMID 24002961
- [Background] Reich KM, Fedorak RN, Madsen K, Kroeker KI. Vitamin D improves inflammatory bowel disease outcomes: basic science and clinical review. World J Gastroenterol. 2014 May 7;20(17):4934-47. doi: 10.3748/wjg.v20.i17.4934. PMID 24803805
- [Background] Romkens TE, van Vugt-van Pinxteren MW, Nagengast FM, van Oijen MG, de Jong DJ. High prevalence of fatigue in inflammatory bowel disease: A case control study. J Crohns Colitis. 2011 Aug;5(4):332-7. doi: 10.1016/j.crohns.2011.02.008. Epub 2011 Mar 24. PMID 21683303
- [Background] Sipponen T, Nuutinen H, Turunen U, Farkkila M. Endoscopic evaluation of Crohn's disease activity: comparison of the CDEIS and the SES-CD. Inflamm Bowel Dis. 2010 Dec;16(12):2131-6. doi: 10.1002/ibd.21300. PMID 20848462
- [Background] Vazquez MA, Lopez E, Montoya MJ, Giner M, Perez-Temprano R, Perez-Cano R. Vertebral fractures in patients with inflammatory bowel disease compared with a healthy population: a prospective case-control study. BMC Gastroenterol. 2012 May 14;12:47. doi: 10.1186/1471-230X-12-47. PMID 22584049